CLINICAL TRIAL: NCT06418191
Title: The Role Of Mobile Applications In Therapy Compliance And Efficacy Of Acupressure In Asthenopia
Brief Title: Mobile Apps Enhancing Acupressure Therapy Compliance and Efficacy for Asthenopia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Dion Rukmindar, Medical Doctor, Indonesia University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-03-0424
Record Dates: First submitted 2024-05-12; First posted 2024-05-17 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Asthenopia
MeSH Terms: conditions — Asthenopia | interventions — Acupressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile app users (Experimental): Mobile application users will be notified twice per day to perform acupressure. Instructions for performing acupressure are in the mobile app
  Interventions: Procedure: Acupressure
- Not a mobile app user (Active Comparator): Non-users of the mobile application will be given an explanation of how to perform acupressure at the start of the study and will not be reminded to perform acupressure therapy.
  Interventions: Procedure: Acupressure

INTERVENTIONS:
Procedure: Acupressure — Acupressure is a technique that involves applying pressure to specific points on the body. It is based on the same principles as acupuncture but uses pressure from fingers, palms, elbows, or specialized devices instead of needles.

SUMMARY:
The goal of this clinical trial is to learn if a mobile application works to improve adherence to acupressure therapy in asthenopia. It will also learn about the efficacy of acupressure as a therapy for asthenopia. The main questions it aims to answer are:

-Does a mobile application have a role to improve therapy compliance and efficacy of self-guided acupressure in asthenopia?

Researchers will compare users of a mobile app to non-users of a mobile app to see if a mobile app works to improve adherence to acupressure therapy in asthenopia

Participants will:

* Do acupressure 2 times every day for 4 weeks
* Filling in the absence link has been after doing acupressure every day
* Fill out the link regarding the condition of asthenopia once per week

DETAILED DESCRIPTION:
This is a clinical trial study to evaluate the role of a mobile application in therapy compliance and acupressure efficacy in asthenopia sufferers. Participants are 60 males/females aged 18-64 years. They will be divided into 2 groups: (1) Acupressure mobile app users and (2) Non-acupressure mobile app users. Acupressure is scheduled 2 times every day for 4 weeks. Therapy compliance will be assessed from the absence link that participants fill out every day, while therapy efficacy will be assessed once per week for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Using a smartphone with the Android platform.
* Work or use digital gadgets for at least 4 hours a day.
* Suffering from asthenopia as indicated by a CVS-Q score ≥ 6.
* Can be contacted with the WhatsApp application.
* Willing to take part in this research until completion and agree to informed consent.

Exclusion Criteria:

* There are tumors, wounds or skin infections in the eye area.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Daily Report of Acupressure | 2 times every day for 4 weeks
  Daily acupressure reports are used to monitor participants' therapeutic compliance in performing acupressure every day

SECONDARY OUTCOMES:
Computer Vision Syndrome Questionnaire (CVS-Q) | Monitored once per week for 4 weeks
  The Computer Vision Syndrome Questionnaire (CVS-Q) is a tool used to assess symptoms related to prolonged computer use or other digital screens. It typically consists of a series of questions designed to evaluate various discomforts experienced by individuals who spend significant time in front of screens. These questions may inquire about symptoms such as eye strain, headaches, blurred vision, dry eyes, neck or shoulder pain, and general fatigue.
  A CVS-Q score ≥ 6 indicates asthenopia
Visual Analog Scale (VAS) | Monitored once per week for 4 weeks
  VAS is used to assess complaints of asthenopia intensity on a scale of 1-10

CONTACTS AND LOCATIONS:
Overall Officials: KEPK FKUI-RSCM, Principal Investigator — The Ethics Committee of the Faculty of Medicine, University of Indonesia - RSCM
Locations (1):
- Cipto Mangunkusumo Hospital, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No